CLINICAL TRIAL: NCT03642496
Title: The Clinical Study of Structurally Optimized ET019002-T Cell Therapy for Refractory/Relapsed B-Cell Malignancies
Brief Title: Clinical Study of ET019002-T Cell Therapy for Refractory/Relapsed B-Cell Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2018LSL-C003
Record Dates: First submitted 2018-08-13; First posted 2018-08-22 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: B-Cell Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- The low dose group (Experimental)
  Interventions: Biological: Low dose ET019002- T Cells
- The middle dose group (Experimental)
  Interventions: Biological: Middle dose ET019002- T Cells
- The high dose group (Experimental)
  Interventions: Biological: High dose ET019002- T Cells

INTERVENTIONS:
Biological: Low dose ET019002- T Cells — ET019002- T Cells are autologous T cells transduced expressing a novel anti-CD19 (ET019002) chimeric antigen receptor,and are administered by intravenous infusion with the dose of 0.75×10*6/kg.
  Arms: The low dose group
Biological: Middle dose ET019002- T Cells — ET019002- T Cells are autologous T cells transduced expressing a novel anti-CD19 (ET019002) chimeric antigen receptor,and are administered by intravenous infusion with the dose of 1.5×10*6/kg.
  Arms: The middle dose group
Biological: High dose ET019002- T Cells — ET019002- T Cells are autologous T cells transduced expressing a novel anti-CD19 (ET019002) chimeric antigen receptor,and are administered by intravenous infusion with the dose of 3.0×10*6/kg.
  Arms: The high dose group

SUMMARY:
This study is to determine the safety, including potential dose limiting toxicities, and efficiency of ET019002-T cells and the duration of in vivo survival of ET019002-T cells in patients with relapsed/refractory B-Cell Malignancies.

DETAILED DESCRIPTION:
ET019002-T cell therapy is a novel chimeric T-cell therapy platform that in preclinical studies, functionally matches the efficacy of CAR-T cells, but dramatically reduces the release of cytokines upon killing of target-positive tumors.The arm of the study is experimental i.v. arm:ET019002-T cells administered by intravenous (IV) infusion.The intervention is ET019002-T cells(Autologous T cells transduced with lentivirus encoding an anti-CD19 (ET019002)-expression construct).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed B cell malignancies including: B-cell Acute Lymphoblastic Leukemia (B-ALL) and B cell lymphomas (DLBCL、FL、MZL、LPL、HCL、CLL、BL、MCL)
* Refractory/Relapsed B cell malignancies:
* Age 6-80 years, male or female
* Nidus could be evaluated: minimum diameter of single nidus ≥10mm, and/or tumor cells in bone marrow ≥ 5%
* ECOG≤2 points
* Function of main organs or tissues were functional: Liver - ALT/AST≤3 normal upper limit, Serum total bilirubin (TBIL) ≤2 normal upper limit; Kidney - glomerular filtration rate (GFR) > 60 mL/min/1.73 m2 or serum creatinine in normal range; Lunge - carbon monoxide diffusion capacity (DLCO) or forced expiratory volume in 1s (FEV) >45% estimate; Heart - left ventricular ejection fraction (LVEF) ≥50%
* Expecting life span ≥3 months
* No chemotherapy, radiation therapy or immunotherapy in 2 weeks before enrollment
* Fertile females/males consented to use contraceptives during participation of the trial
* Patient or his/her custodia could understand and is willing to sign the written consent

Exclusion Criteria:

* Pregnancy or lactation
* Couldn't use contraceptives during participation of the trial
* Couldn't collect enough monocyte
* Active and/or severe infection
* HIV infection, active Hepatitis B or Hepatitis C infection
* Had active autoimmune disease
* Had non-melanoma skin carcinoma (NMSC) or Carcinoma in situ (e.g. cervix, bladder, galactophore)
* Obvious clinical encephalopathy or novel neuron function damage
* Organ failure: Heart - upper than NYHA level III or had uncontrolled malignant arrhythmia; Liver - upper than level III of Wuhan conference classification; Kidney - kidney failure stage3 or worse
* Using immunosuppressive drugs or adreno-cortical hormone (ACH) within two weeks of enrollment
* Insufficient T cell number or T cell transfection rate
* Needed urgent disease controlling due to tumor load
* Patients had biological treatment, immunotherapy or radiation therapy within 6 weeks prior to enrollment or are currently under these treatment
* Substance abuse or drug addiction
* lack of compliance, communication deficit or other unaccommodated situations

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-08-19 (Estimated); Primary Completion 2020-08-19 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 12 weeks.
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the ET019002T-cells,which is irreversible or life threatening or CTCAE Grade 3-5.
Tmax of serum cytokine levels | Up to 12 weeks.
  Cytokins as measured by CBA-Bioplex Multiplex Immunoassays will be presented as time to peak level.
Time to baseline for serum cytokine levels | Up to 12 weeks.
  Inceases or decreases in the amout of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing.
Toxicity profile of ET019002T-cell treatment | Up to 2 years.
  Frequency of treatment-related adverse events that occurred at any time from the first day of infusion that are "possibly", "likely", or "definitely" related to the study, including infusion related toxicity and ET019002 T cell related toxicity. Include but not limited to: Fever, chills, nausea, vomiting, jaundice and other gastrointestinal symptoms; Fatigue, hypotension, respiratory distress; Tumor lysis syndrome; Cytokine release syndrome; Neutropenia, thrombocytopenia; Liver and kidney dysfunction. Assessed at all visits.

SECONDARY OUTCOMES:
Rate of disease response | Up to 12 weeks.
  Rate of disease response assessed by lugano cliassification.Response rates will be estimated as CR,PR,SD,PD.
Progression free survival(PFS) | Up to 2 years.
  Progression free survival(PFS) denotes the chances of staying free of disease progression for patients after treatment.
Time to baseline for B cell level | Up to 2 years.
  B cell level as measured by Bio-Plex Multiplex Immunoassays will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: He Peng cheng, Doctor, Principal Investigator — First Affiliated Hospital of Xian JiaotongUniversity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He P, Liu H, Zimdahl B, Wang J, Luo M, Chang Q, Tian F, Ni F, Yu D, Liu H, Chen L, Wang H, Zhang M, Grupp SA, Liu C. A novel antibody-TCR (AbTCR) T-cell therapy is safe and effective against CD19-positive relapsed/refractory B-cell lymphoma. J Cancer Res Clin Oncol. 2023 Jul;149(7):2757-2769. doi: 10.1007/s00432-022-04132-9. Epub 2022 Jul 1. PMID 35776199